CLINICAL TRIAL: NCT01909843
Title: A Phase I, Single-centre, Open Label Study to Evaluate the Potential Occurrence, Reversibility and Prevention of Bronchoconstriction as Individual Response to Escalating Doses Followed by Repeated Doses of ALX-0171, Administered by Oral Inhalation to Adults With Hyperresponsive Airways
Brief Title: ALX-0171 Safety Study in Adults With Hyperresponsive Airways
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALX-0171-1.2/13; 2012-005811-14 (EudraCT Number)
Record Dates: First submitted 2013-07-24; First posted 2013-07-29 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Respiratory Syncytial Virus Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — gontivimab

ARMS (1):
- ALX-0171 Oral inhalation (Experimental)
  Interventions: Biological: ALX-0171

INTERVENTIONS:
Biological: ALX-0171 — Escalating dose of ALX-0171 during maximum 3 consecutive days: from 2.1 mg to maximum 200 mg per inhaled dose followed by daily dose of 70 mg, 140 mg or 200 mg per dose for maximum 4 consecutive days

SUMMARY:
This is a Phase I, single-centre, open label study to evaluate the occurrence and subsequent reversibility and prevention, of bronchoconstriction following single and repeated oral inhalations of ALX-0171 in adults with hyperresponsive airways.

This phase I study is an exploratory study and serves to evaluate the occurrence and reversibility of bronchoconstriction upon inhalation of ALX-0171. The study is an open label trial with a sequential administration regimen of placebo and verum in all planned study subjects. Each subject will start the treatment with a single dose of ALX-0171 placebo (= formulation buffer) followed by escalating doses of ALX-0171 verum.

Eventually a second administration of ALX-0171 placebo may take place at the end of the study (as defined per protocol).

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female subjects aged 18-60 years (both included).
2. Subjects must demonstrate a PC20 (concentration of the agonist in the inhaled substance leading to a fall in FEV1 of ≥20.0% of personal best at same visit) response to methacholine (MCh) concentrations of > 1 mg/mL and ≤ 8 mg/mL at screening.
3. Subjects not on concomitant treatments except for

   1. medication that has no effect on hyperresponsiveness, bronchoconstriction or on lung function parameters
   2. respiratory medication for which subjects are able to discontinue their current treatment during the study period taking into account the respective wash-out periods as listed in the protocol.
   3. short-acting bronchodilators under certain conditions as specified in the protocol.
4. Screening forced expiratory volume (FEV1) value of > 60.0% of the predicted normal value after a wash-out of respiratory medication as listed in the protocol.
5. Subject has been informed both verbally and in writing about the objectives of the clinical trial, the methods, the anticipated benefits and potential risks and the discomfort to which he may be exposed, and has given written consent to participation in the trial prior to trial start and any trial-related procedure.
6. Body weight according to a Body Mass Index ≥ 18.5 and ≤ 29.0 kg/m².
7. Non-smokers or ex-smokers who have stopped smoking for at least 1 year prior to start of the clinical study. No history of smoking more than 10 pack years.
8. Ability to inhale in an appropriate manner.
9. Female subjects of childbearing potential and male subjects must agree to use appropriate methods of contraception as specified in the protocol.

Exclusion Criteria:

1. Subjects with a pre-dose baseline FEV1 measurement on the first day (i.e. prior to the first inhalation of ALX-0171 placebo) which is below or equal to 60.0% of the predicted FEV1 value.
2. Presence of clinically significant diseases other than asthma, hyperresponsive airways or atopic diseases (cardiovascular, renal, hepatic, gastrointestinal, haematological, neurological, genitourinary, autoimmune, endocrine, metabolic, etc.), which, in the opinion of the investigator, may either put the subject at risk because of participation in the trial, or diseases which may influence the results of the study or the subject's ability to take part in it.
3. Presence of relevant pulmonary diseases (except asthma) or history of thoracic surgery.
4. History or current evidence of clinically relevant allergies to drugs.
5. Any absolute or relative contraindications for methacholine challenge: e.g., severe or moderate airflow limitation (FEV1 ≤ 60.0% predicted or < 1.5 L), heart attack or stroke in the last 3 months, uncontrolled hypertension, known aortic aneurysm, current use of cholinesterase inhibitor medication.
6. Hospitalisation or emergency room treatment for acute asthma in the 3 months prior to screening, between screening and the start of the treatment period.
7. Hospitalisation for longer than 24 hours for the management of an asthma exacerbation within the preceding 3 months of the screening visit or intubation (ever) for that named cause.
8. History of allergic reactions to any active or inactive ingredients of the nebuliser solution.
9. ECG abnormalities of clinical relevance.
10. Clinically relevant abnormal heart rate and/or blood pressure as judged by the investigator.
11. Proneness to orthostatic dysregulation, fainting, or blackouts.
12. History (within the last 5 years) or presence of any malignancy except for basalioma.
13. Clinically relevant abnormalities in clinical chemical, haematological or in any other laboratory variables.
14. Chronic or clinically relevant acute infections.
15. Clinically relevant positive results in any of the following virology tests: Hepatitis B surface antigen, Hepatitis C antibodies, human immunodeficiency virus (HIV)-1, and HIV -2 antibodies.
16. Positive drug screen.
17. History of previous administration of ALX-0171 or any other medication targeting the F-protein (e.g. palivizumab) or any other inhaled biologic. In any other case of use of biologics: 6 months, or the time of duration of the pharmacodynamic effect, or 10 times the half-life of the respective drug, whatever is longer, before first trial medication administration.
18. History or presence of alcohol or drug abuse.
19. Planned donation of germ cells, blood, organs, bone marrow during the course of the trial or within 6 months thereafter.
20. Participation in another clinical trial with an investigational drug within the last month (defined as 1 month between last visit previous trial and Informed Consent Form (ICF)signature of the current trial).
21. Blood donation within the last 30 days before screening.
22. Lack of ability or willingness to give informed consent.
23. Anticipated non-availability for trial visits/procedures.
24. Anticipated lack of willingness or inability to cooperate adequately.
25. Vulnerable subjects (e.g., persons kept in detention).
26. Consumption of any xanthine derivates (such as -but not limited to-, caffeine, theophylline, chocolate) 6 hours before first procedure at each study visit.
27. Pregnant or lactating women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects reacting with bronchoconstriction to treatment (ALX- 0171 placebo or ALX-0171 verum) with one or more drops in forced expiratory volume in one second (FEV1) within a period of 8h post-inhalation | Within a period of 8 hours post-inhalation

SECONDARY OUTCOMES:
Total number of bronchoconstriction events | Day 1 to Day 7
The frequency of use of β2-agonist for the treatment of study drug/procedure induced bronchoconstriction | Day 1 to Day 7
Safety markers | From screening to last follow-up visit which will take place between day 35 and day 42
  between others: physical examination, vital signs, 12-lead ECG, clinical laboratory (hematology and serum chemistry), urine analysis, serology, adverse events
Pharmacokinetic parameters: plasma concentrations of ALX-0171 | Day 1 to Day 8
Immunogenicity: presence of anti-drug antibodies (ADA) in serum, presence of ADA in sputum | From screening to last follow-up visit which will take place between day 35 and day 42

CONTACTS AND LOCATIONS:
Overall Officials: Steven De Bruyn, MD, Study Director — Ablynx NV
Locations (1):
- Gauting, Germany